CLINICAL TRIAL: NCT07056452
Title: Hydrodissection Circumcision Versus Conventional Circumcision: A Randomized Trial Evaluating Efficacy, Safety, and Patient Outcomes in Male Circumcision
Brief Title: Hydrodissection Circumcision Versus Conventional Circumcision
Acronym: Circumcision
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Collaborators: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Wujiang Liu, Professor, Peking University
Other Study IDs: CQJLPWCH-008; 510212197105014555 (Registry Identifier: Liu Wujiang)
Record Dates: First submitted 2025-03-09; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-03

CONDITIONS: Circumcision
Keywords: Circumcision; Hydrodissection; HC; sCC; uCC

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm 1: Control Group: This group has not hydrodissection but has tissue sparing
- Arm2: Control Group: This group has not hydrodissection and also hasn't tissue sparing
- Arm3: Hydrodissection circumcision: By injecting a solution of physiological saline containing 0.5% lidocaine along the cutting line , the hydrodissection technique creates a natural plane of separation, facilitating precise and minimally invasive skin removal.
  Interventions: Procedure: hydrodissection technique

INTERVENTIONS:
Procedure: hydrodissection technique — injecting a solution of physiological saline containing 0.5% lidocaine along the cutting line
  Groups: Arm3: Hydrodissection circumcision

SUMMARY:
Over a period of more than 3 years (January 2021 to February 2024), 96 males (aged 6-35 years; average 12.3 years) who underwent circumcision were randomly divided into three groups: HC, sCC (tissue sparing), and uCC (tissue unsparing), with a follow-up period exceeding 1 year.

The HC group used physiological saline containing 0.5% lidocaine for hydrodissection, while the CC group did not have a hydrodissection step.

Outcome Measurements and Statistical Analysis: Primary outcomes: operation time, intraoperative bleeding, postoperative pain and wound healing time. Secondary outcomes: intraoperative pain, postoperative complications and cosmetic results. The statistical analysis of results follows the randomized case-control trial (RCT) analysis method.

DETAILED DESCRIPTION:
Participants were randomized 1:1:1 to the hydrodissection or conventional group using computer-generated random numbers. Surgeons and patients were blinded to group allocation until the procedure began. Based on the previous research results, with reference to the mean and standard deviation range, the sample size is calculated to be at least 28 cases per group (α=0.05, β=0.2). Considering the proportion of lost to follow-up, we selected 32 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* Complies with the diagnostic criteria for phimosis, foreskin elongation, and related diseases in the "Chinese Expert Consensus on Phimosis, Foreskin related Diseases";
* Preoperative routine examination showed no abnormalities in coagulation, blood routine, electrocardiogram and other indicators;
* No severe genital herpes, gonorrhea, syphilis, glans infection, etc.;
* Complies with the indications for sleeve type circumcision ;
* The patient or family member is aware of the surgical plan and signs the informed consent form.

Exclusion Criteria:

* Patients with concomitant urethral malformations, such as hypospadias;
* Patients with combined inflammation of the penis, prior penile surgery, severe adhesions, buried penis, and short frenulum of the penis;
* Exclude individuals with combined allergies or allergies to multiple medications;
* Patients with severe physical illnesses such as heart and lung dysfunction who cannot tolerate surgery;
* Individuals with cognitive impairments or mental abnormalities;
* Diabetes with poor glycemic control；
* Age >35 or Age<6.

Ages: 6 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — male
Study Population: Outpatient patient requests circumcision
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
operation time | 1 day
  Operative time was calculated by timer.
intraoperative bleeding | 1 day
  The amount of intraoperative bleeding is calculated by weighing gauze before and after operation. 1 milliliter is approximately equal to the weight of 1 gram.
The healing time | 7-25 days
  The healing time was judged by the doctors based on the observation of the wound and inquiry of the patients during 7-25 days after surgery. We defined complete wound healing as the absence of a scab with a completely epithelialized and dry skin surface based on clinical assessment
Intra-operative pain | 1 day
  Intra-operative pain was graded immediately after the operation while the post-operation pain was graded at 1 week by NRS (Numeric Rating Scale). The scale typically ranges from 0 to 10. 0 indicates no pain, while 10 signifies the most severe pain imaginable.

SECONDARY OUTCOMES:
other complications | through study completion, an average of 1 year
  incidence rate
patient satisfaction | through study completion, an average of 1 year
  Patient satisfaction is divided into 5 levels：Extremely dissatisfied，Dissatisfied，Neutral，Satisfied，Extremely Satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Wujiang Liu, Principal Investigator — Peking University
Locations (2):
- China (2):
  - Deparment of Urology, Peking University First Hospital, Beijing, Beijing Municipality
  - Chongqing Jiulongpo District Maternal and Child Health Hospital, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: Yes
All follow up data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after publication
Access Criteria: All interested doctors, professors, and scholars
URL: https://batcmd.com/windows/10/services/dssvc/

DOCUMENTS (1):
  • Study Protocol (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT07056452/Prot_000.pdf